CLINICAL TRIAL: NCT06727669
Title: Longitudinal Cohort of Thrombosis and Hemostasis Diseases
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice President of Peking University Institute of Hematology Affiliation: Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: 2024PHB401-001
Record Dates: First submitted 2024-12-02; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Immune Thrombocytopenia; Thrombotic Thrombocytopenic Purpura; Hemophilia A, Acquired; Disseminated Intravascular Coagulation; Thrombophilia; Deep Vein Thrombosis; Pulmonary Embolism; Thrombotic Microangiopathies; Coagulation Factor Deficiency; Hemophilia A; Hemophilia B; Hemophilia B, Acquired; Platelet Dysfunction; Arterial Thromboembolism; Bleeding Disorder; Thrombosis
Keywords: Thrombosis; Hemostasis
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombotic Thrombocytopenic; Factor 8 deficiency, acquired; Disseminated Intravascular Coagulation; Thrombophilia; Venous Thrombosis; Pulmonary Embolism; Thrombotic Microangiopathies; Hemophilia A; Hemophilia B; Hemostatic Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, prospective, longitudinal, observational cohort study to investigate thrombosis and hemostasis diseases in Chinese patients. This study will collect basic information, diagnostic and treatment information, as well as medical expense information of patients from medical records.The incidence and risk factors of thrombosis and hemostasis diseases, the treatment methods, prognosis and medical expenses of these patients in China will be analyzed. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

DETAILED DESCRIPTION:
Thrombosis and hemostasis diseases are a group of high-risk hematological diseases, characterized by bleeding or hypercoagulability caused by congenital or acquired abnormalities in hemostasis, coagulation, and fibrinolysis. Thrombosis and hemostasis diseases included various bleeding and thrombotic diseases such as primary immune thrombocytopenia (ITP), thrombotic thrombocytopenic purpura (TTP), hemophilia, disseminated intravascular coagulation (DIC), thrombophilia, pregnancy with ITP, pregnancy with prethrombotic state (such as protein C, protein S deficiency, etc.), deep vein thrombosis, pulmonary embolism, thrombocytopenia and coagulation abnormalities after hematopoietic stem cell transplantation, and so on. Thrombosis and hemostasis diseases have a high incidence rate, may affect patients' quality of life and even are associated with the poor survival. However, current studies are mostly based on data from limited sample size cohorts, lacking comprehensive and large-scale prospective cohort studies.

This is a multicenter, prospective, longitudinal, observational cohort study investigating the incidence and risk factors of thrombosis and hemostasis diseases, and to analyze the treatment methods, prognosis and medical expenses of these patients in China.This study will collect basic information, diagnostic and treatment information, as well as medical expense information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as thrombosis and hemostasis diseases.

Exclusion Criteria:

* Long-term follow-up information for patients is not available for any reason, such as not being available or having a serious concomitant disease.
* Patients with alcohol and drug addictions or mental illness affect their ability to comply with study requirements.
* According to the investigator, there are conditions that may endanger the patient's safety or affect his/her compliance.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed as thrombosis and hemostasis diseases, including immune thrombocytopenia, thrombotic thrombocytopenic purpura, hereditary and acquired Hemophilia, disseminated intravascular coagulation, pregnancy With ITP, pregnancy With prethrombotic state (such as protein C, protein S deficiency, etc.), deep vein thrombosis, pulmonary embolism, thrombocytopenia and coagulation abnormalities after hematopoietic stem cell transplantation, hereditary and acquired thrombophilia,hereditary hemorrhagic disease , et al.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognosis | 5 years
  To analyze the long-term prognosis of patients with thrombosis and hemostasis diseases, such as immune thrombocytopenia (ITP),thrombotic thrombocytopenic purpura, hereditary and acquired hemophilia, disseminated intravascular coagulation, pregnancy With ITP, pregnancy With prethrombotic state (such as protein C, protein S deficiency, etc.), deep vein thrombosis, pulmonary embolism, thrombotic microangiopathies, thrombocytopenia or coagulation abnormalities after hematopoietic stem cell transplantation, hereditary and acquired thrombophilia, platelet dysfunction,arterial thromboembolism, and hereditary hemorrhagic disease , et al., and analyze the risk factors associated with their prognosis.

SECONDARY OUTCOMES:
Incidence | 5 years
  To describe the incidence of thrombosis and hemostasis diseases, and analyze the risk factors associated with these diseases.
Distribution | 5 years
  The population characteristics of thrombosis and hemostasis diseases
Overall response rate | 180 days
  To analyze the therapeutic efficacy of patients with thrombosis and hemostasis diseases, and analyze the impact factors associated with the efficacy.
Long-term overall remission rate | 1 years
  Proportion of the participants with an overall remission.
Safety of treatment | 1 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Health economic evaluation | 5 years
  To perform hospital stay and hospitalization cost evaluation in patients with thrombosis and hemostasis diseases

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (5):
- China (5):
  - Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality
  - Department of Hematology, Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Department of Hematology, Beijing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xinqiao Hospital, Army Military Medical University, Chongqing